CLINICAL TRIAL: NCT03407950
Title: Cognitive Remediation Program for Hospitalized in the Long Term Patients With Deficit Schizophrenia : Impact on the Capacities of Autonomy
Brief Title: Cognitive Remediation Program for Hospitalized in the Long Term Patients With Deficit Schizophrenia
Acronym: IPT+
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study stopped due to major feasibility issues and the notices was expired.
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9529
Record Dates: First submitted 2017-11-14; First posted 2018-01-23 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Schizophrenia
Keywords: Deficit Schizophrenia; long stay inpatients; cognitive remediation; negative symptoms
MeSH Terms: conditions — Schizophrenia | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group IPT+ (Other): 2 sessions of IPT+ by week during 6 months
  Interventions: Behavioral: IPT+
- Control Group (Other): group without specific therapy (Treatment as usual) but same number and duration of each sessions than IPT+
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: IPT+ — Integrated Psychological Treatment and cognitive remediation and relaxation and Mindfulness : IPT+. A blind evaluation will be realized thanks to questionnaires of the current practice to compare the IPT+ versus treatment as usual (TAU).
  Arms: Group IPT+
Behavioral: Treatment as usual — no specific therapy but same number and duration of each sessions than IPT+. A blind evaluation will be realized thanks to questionnaires of the current practice to compare the IPT+ versus treatment as usual (TAU).
  Arms: Control Group

SUMMARY:
Schizophrenia is a chronic disease with deficit in social interaction and lost of autonomy in daily life. Negative symptoms as blunted affect, avolition, social deficit and anhedonia and cognition were prognosis and functioning key's factors. Psychotropic medications have shown only poor effect to improve negative symptoms and cognition as attention, memory and cognitive flexibility. So, cognitive remediation programs were developped to focus cognitive disorders. The IPT (Integrated Psychological Treatment) is one of the most complete program with modules on cognitive and social abilities. The aim of this study is to evaluate the efficacy of IPT+ program to improve autonomy capacities of long stay inpatients suffering from schizophrenia 6 at the end of the program With IPT+ this study will improve autonomy capacities for patients suffering from deficit schizophrenia and allowed patients to go out hospital earlier than before.

DETAILED DESCRIPTION:
Schizophrenia is a chronic disease with deficit in social interaction and lost of autonomy in daily life. Negative symptoms as blunted affect, avolition, social deficit and anhedonia and cognition were prognosis and functioning key's factors. Psychotropic medications have shown only poor effect to improve negative symptoms and cognition as attention, memory and cognitive flexibility. So, cognitive remediation programs were developped to focus cognitive disorders. The IPT (Integrated Psychological Treatment) is one of the most complete program with modules on cognitive and social abilities. The aim of this study is to evaluate the efficacy of IPT+ program to improve autonomy capacities of long stay inpatients suffering from schizophrenia 6 at the end of the program The secondary objectives are to evaluate autonomy 6 months after the program, to evaluate the efficacy of the program on negative symptoms, quality of life, cognitive functions, social cognition and duration of hospitalisation.

This study propose a randomised controlled study with 2 arms, with blind evaluation to compare the IPT+ versus treatment as usual (TAU). The follow up will be 6 month for the With IPT+ this study will improve autonomy capacities for patients suffering from deficit schizophrenia and allowed patients to go out hospital earlier than before.

ELIGIBILITY:
Inclusion criteria:

* age > 18 and < 60
* Diagnosis of schizophrenia on DSM 5
* criteria of deficit schizophrenia with the schedule for deficit syndrome
* inpatient at inclusion with at least 6 month of hospitalisation during the last 2 years
* clinically stable
* able to understand, talk and read french
* signing consent form

Exclusion criteria:

* change in psychotropic treatment during the last month
* psychotherapy in the last 8 months or planned during the study
* CDSS score > 9
* drug dependency during the last year
* unstable somatic disease
* somatic disease with impact on cognition

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Social autonomy | 6 months
  Evaluated by Social autonomy Scale (EAS). It's a scale composing by 17 highly-rated items from 0 to 6 (total score varying 0 in 102, a low score indicating a better social autonomy).

SECONDARY OUTCOMES:
Clinical symptomatology | 6 and 12 months
  Evaluated by the Assessment of Negative Symptoms (SANS). It's a scale composing by 25 items, highly-rated from 0 to 5.
Clinical symptomatology | 6 and 12 months
  Evaluated by the Lille Apathy Rating Scale (LARS). It's a scale composing by 33 questions distributed in 9 columns. A global score is calculated varying of "36-22" (No apathetic person), "21-17" (trend to the apathy), "-16 in -10" (Moderate apathy) and of "-9 has + 36" (Severe apathy).
Clinical symptomatology | 6 and 12 months
  Evaluated by the Social Anhedonia Scale (SAS). It's a scale composing by 40 items quoted by the subject in "truth" or "false".
Clinical cognition | 6 and 12 months
  Evaluated by scale D2 test
Clinical cognition | 6 and 12 months
  Evaluated by scale Trail Making Test (TMT)
Clinical cognition | 6 and 12 months
  Evaluated by scale California Verbal Learning Test (CVLT)
Clinical cognition | 6 and 12 months
  Evaluated by scale WAIS III. The total score varies between 0 and 21
Clinical cognition | 6 and 12 months
  Evaluated by scale ER-40. It's an computer-based testing translates into French and which lasts 6 minutes. It consists with 40 photos of faces expressing 4 basic feelings (enjoyment, sadness, anger and fear) or neutrals. In every thrown image, 5 choices of feelings are possible.
Clinical cognition | 6 and 12 months
  Evaluated by Social cognition. A score of global social support will be estimated, between 0 (no knowledge, no possibility of emotional or financial support by other people) and 5 (patient having the possibility of living or living at a close person, anybody () gets fresh ideas worrying about the patient and about his coverage(care) and suggesting accompanying him(it) in the diverse administrative procedures or with care, very supported and varied emotional circle of acquaintances, possible financial support by the close friends(relations) and the guarantor(respondent) entirely for the necessities of the patient).
Clinical cognition | 6 and 12 months
  Evaluated by scale to assess Unawareness of Mental Disorder (SUMD). The answers are quoted(esteemed) from 1 to 5. The highest scores indicate the highest levels of non-consciousness of the disorder.
Clinical functioning | 6 and 12 months
  Evaluated by scales Quality of life (S-QoL-18)
Clinical functioning | 6 and 12 months
  Evaluated by scale Warwick-Edinburgh Mental Well-Being Scale (WEMWBS). Items are quoted of 1 (never) in 5 (all the time) giving a total score between 14 and 70.
Clinical functioning | 6 and 12 months
  Evaluated by scale Emotional Reactivity Scale (ERS). The 13 items are quoted of 0 (never) in 4 (always).

CONTACTS AND LOCATIONS:
Overall Officials: Delphine CAPDEVIELLE, PU-PH, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Delphine CAPDEVIELLE, Montpellier, France

IPD SHARING:
Plan to Share IPD: No